CLINICAL TRIAL: NCT05830097
Title: An Open-Label, Non-randomized, Multinational, Multi-center Phase I/Ⅱ Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Bi-Ligand-Drug Conjugate CBP-1019 in Patients With Advanced Solid Tumors
Brief Title: A Study of Bi-Ligand-Drug Conjugate CBP-1019 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coherent Biopharma (Hefei) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP-1019-101
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2023-12

CONDITIONS: Cancer, Breast; Cancer, Lung; Cancer of Pancreas; Cancer of Esophagus; Cancer Colorectal
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Colonic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ia stage - CBP-1019 Dose escalation/ Ib、II stage - CBP-1019 monotherapy (Experimental): Ia:Patients will receive CBP-1019 IV infusion every 2 weeks until disease progression, intolerability, informed consent withdraw, or other reasons leading to treatment discontinue.
  Ib:Patients will receive CBP-1019 RP2D IV infusion every two weeks until disease Patients will receive CBP-1019 RP2D IV infusion every two weeks until disease progression, intolerability, informed consent withdraw, or other reasons leading to treatment discontinue.
  Interventions: Drug: CBP-1019

INTERVENTIONS:
Drug: CBP-1019 — Light yellow to yellow loose lumps or powder；50mg/vial; Infusion for 90 minutes (± 10 minutes), once every 2 weeks.
  Other Names: CBP-1019 for injection

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and potential efficacy and to determine the recommended phase 2 dose (RP2D) of CBP-1019, a bi-specific ligand conjugated drugs in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This phase Ia and Ib/II, open-label, multicenter study has two stages. The Ia stage is a dose-escalation study that will focus on safety, tolerability, pharmacokinetics, maximum tolerated dose (MTD) and phase 2 dose (RP2D). Patients with advanced solid tumor who failed from previous standard treatment or without standard therapy exists will be enrolled in the phase Ia study. Dose-limiting toxicity (DLT) observation period is 28 days.

Patients in phase Ib/II part will be recruited into certain tumor cohorts and receive RP2D CBP-1019 iv infusion every two weeks. Primary efficacy of objective response rate (ORR), disease control rate (DCR), progression free survival (PFS), etc., will be evaluated. The correlation between tumor response and the receptors will be explored. Safety information will be collected in phase Ib/II stage.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent form (ICF) prior to any study-specific procedures.
2. Men or women ≥ 18 years old when signed ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS)0-1
4. Life expectancy of ≥ 3 months, in the opinion of the Investigator.
5. Pathologically documented advanced solid tumor, including but not limited to advanced lung cancer, pancreatic cancer, colorectal cancer, esophageal cancer, and breast cancer, etc.
6. The tumor tissue should be provided for folate receptor α (FRα) and transient receptor potential cation channel subfamily V member 6 (TRPV6) immunohistochemistry (IHC) testing, optional for low dose level (≤ 2.0 mg/kg) of phaseⅠa. Tumor FRα and TRPV6 expression as determined by an IHC assay performed by a central laboratory on previously obtained archival tumor tissue or tissue obtained from a biopsy at screening.
7. Subjects must have received prior standard therapy appropriate for their tumor type and stage of disease, or in the opinion of the investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy, or absence of standard therapy.
8. Progress of disease per response evaluation criteria in solid tumors (RECIST) 1.1 after the last anti-tumor treatment (solid tumors).
9. At least one measurable soft tissue lesion per RECIST 1.1, lesions received prior radiotherapy can be regarded as measurable only when occurring conclusive progression after radiotherapy, optional for low dose level (≤ 2.0 mg/kg) of Phase Ⅰa.
10. Adequate bone marrow and organ function, defined as:

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
    * Platelet count ≥ 100 × 109/L.
    * Hemoglobin (Hb) ≥ 90 g/L.
    * Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), or ≤ 2 × ULN for subjects with liver metastases.
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN, or ≤ 2 × ULN for subjects with liver metastases.
    * Creatinine clearance (CCr) ≥ 60 mL/min as calculated using Cockcroft-Gault formula
11. Women of child-bearing potential (WOCBP) or male subjects whose spouse is WOCBP need to adopt a medically approved contraceptive measure (such as intra-uterine device (IUD), contraceptive pill, or condom) throughout the study and for at least 3 months in males and 6 months in females after the last dose of CBP-1019.

Exclusion Criteria:

1. Known prior or suspected hypersensitivity to CBP-1019 or any component in their formulations.
2. Concurrent malignancy within 5 years prior to the first dose of CBP-1019, other than clinically considered cured early malignant tumors (carcinoma in situ or stage I tumor) such as basal cell carcinoma, localized squamous cell cancer of the skin, Superficial bladder cancer, etc.
3. Central nervous system (CNS) metastasis and/or carcinomatous meningitis. Treated CNS metastasis may be enrolled only if it is stable for at least 1 month, no evidence of new or expanded lesions exist, and steroid treatment has been discontinued at least 3 days before the first dose of CBP-1019.
4. Poorly controlled pleural effusion, pericardial effusion, or ascites, or those need repeated drainage, such as drainage once a month or more frequently, or within 2 weeks before the dose of CBP-1019.
5. Washout periods of prior anti-tumor treatments have not been completed.
6. Any toxicities of prior anti-cancer therapy not resolved to Grade 1 per NCI CTCAE 5.0 or inclusion criteria, other than alopecia and fatigue.
7. Fever >38.5 °C of unknown cause.
8. Positive Hepatitis B Surface Antigen (HbsAg) and Hepatitis B virus (HBV) DNA ≥ 500 IU/mL or 2500 copies or lower limits of normal (LLN) of positive.
9. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).

10 History of clinically significant vascular diseases, including acute arteriovenous embolism, acute thrombotic arteritis, thrombophlebitis, acute pulmonary embolism, acute coronary syndrome .

11. History of treated active gastrointestinal ulcers, perforations, and/or fistulas within 6 months prior to the first dose of CBP-1019.

12. History of autoimmune disease, immunodeficiency disease and organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | up to 12 months
  Safety and tolerability: incidence of dose limiting toxicities (DLTs)、treatment emergent adverse events、serious adverse events (SAEs)、electrocardiogram (ECG) and clinical laboratory tests per the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE 5.0).

SECONDARY OUTCOMES:
MTD/RP2D of CBP-1019. | Up to 28 days after the first dose of CBP-1019
  Dose limiting toxicity (DLT) will be assessed by NCI CTCAE v5.0.Critical decisions as DLT/MTD/RP2D evaluation and dose escalation will be made by Safety monitoring committee (SMC).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (5):
- United States (4):
  - TOI Clinical Research LLC, Cerritos, California
  - Florida Cancer Specialists & Research Institute, Orlando, Florida
  - Northwell Health Inc., Manhasset, New York
  - Next Oncology, Fairfax, Virginia
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No